CLINICAL TRIAL: NCT02108483
Title: Phototoxicity Test of Dapsone Gel in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 225678-010
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): Dapsone gel and dapsone gel vehicle applied to the skin by separate occlusive patches on Day 1.
  Interventions: Drug: dapsone gel; Drug: dapsone gel vehicle

INTERVENTIONS:
Drug: dapsone gel — Patches containing dapsone gel will be applied to the skin.
Drug: dapsone gel vehicle — Patches containing dapsone gel vehicle will be applied to the skin.

SUMMARY:
This study will evaluate the potential of dapsone gel and its vehicle to cause a phototoxic reaction following irradiation of the skin under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

-Healthy adults.

Exclusion Criteria:

* Skin diseases, excessive hair, tattoos, pigmentation, scars or moles that could interfere with patch application
* Sensitivity to adhesive bandages or tape.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Phototoxicity Irritation Potential Using a Visual Scale | 4 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fair Lawn, New Jersey, United States